CLINICAL TRIAL: NCT05258474
Title: A Phase I, Double-blind, Randomised, Placebo-controlled, Single-ascending and Multiple-ascending Dose Trial to Evaluate Safety and Pharmacokinetics of Oral Controlled-ileocolonic-release Nicotinamide (CICR-NAM) Compared to Immediate-release Nicotinamide and Placebo in Healthy Subjects and in Patients With Inflammatory Bowel Diseases
Brief Title: Safety and Pharmacokinetics of Oral Controlled-ileocolonic-release Nicotinamide (CICR-NAM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CICR-NAM; 2020-002815-23 (EudraCT Number); DRKS00023384 (Registry Identifier: DRKS - German Clinical Trials Register)
Record Dates: First submitted 2021-08-19; First posted 2022-02-28 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Safety Issues; Pharmacokinetic
Keywords: Nicotinamide; Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Sagittal Abdominal Diameter

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- healthy subjects (Experimental): healthy subjects (single-ascending and multiple-ascending doses)
  Interventions: Drug: controlled-ileocolonic-release nicotinamide (SAD/MAD/MD); Drug: Immediate-release nicotinamide (SAD); Drug: Placebo controlled-ileocolonic-release nicotinamide (SAD/MAD); Drug: Placebo Immediate-release nicotinamide (SAD)
- IBD-patients (Experimental): inflammatory bowel disease patients (multiple dose)
  Interventions: Drug: controlled-ileocolonic-release nicotinamide (SAD/MAD/MD)

INTERVENTIONS:
Drug: controlled-ileocolonic-release nicotinamide (SAD/MAD/MD) — single- and multiple-ascending dose (SAD/MAD) or multiple dose (MD)
  Other Names: CICR-NAM (SAD/MAD/MD)
Drug: Immediate-release nicotinamide (SAD) — single-ascending dose (SAD)
  Other Names: ImR-NAM (SAD)
  Arms: healthy subjects
Drug: Placebo controlled-ileocolonic-release nicotinamide (SAD/MAD) — single- and multiple-ascending dose (SAD/MAD)
  Other Names: no active substance
  Arms: healthy subjects
Drug: Placebo Immediate-release nicotinamide (SAD) — single-ascending dose (SAD)
  Other Names: no active substance
  Arms: healthy subjects

SUMMARY:
Double-blind, randomised, placebo-controlled phase I trial with single-ascending and multiple-ascending dose to evaluate safety and pharmacokinetics of oral controlled-ileocolonic-release nicotinamide (CICR-NAM) compared to immediate-release nicotinamide and placebo in healthy subjects and in patients with inflammatory bowel diseases.

DETAILED DESCRIPTION:
Nicotinamide (NAM) has been implicated in the restoration and maintenance of a healthy gut microbiome. Conventional NAM formulations are designed for systemic NAM supplementation and therefore release NAM in the stomach and upper small intestine for maximum absorption. In contrast, the novel CICR-NAM tablets (controlled-ileocolonic-release nicotinamide) start releasing in the lower small intestine for topical delivery of NAM to the microbiota and the mucosa in the ileum and colon, also leading to a reduced systemic exposure. This clinical Phase I trial investigates the safety and tolerability of CICR-NAM in single- and multiple-ascending doses (1, 2 and 4 g). At the beginning of the trial, single-dose pharmacokinetics (PK) of 1 g of conventional immediate-release NAM and CICR-NAM are compared. At the end of the trial, patients with inflammatory bowel diseases (IBD) receive a medium multiple dose (2 g for 4 weeks) to compare their exposure, PK and safety data with those of healthy subjects at the same dose level.

ELIGIBILITY:
Main inclusion and exclusion criteria

Inclusion criteria for the SAD and MAD parts with healthy subjects:

1. Male and female subjects aged 18 to 75 years.
2. Healthy subjects without relevant medical conditions.
3. Ability to understand and comply with the protocol.
4. Signed written Informed Consent.
5. A BMI of 18.5 to 29.99 kg/m².
6. Non-smoker or light smoker (average of <7 cigarettes per week) and no history of longterm, heavy smoking (>10 pack-years).

Inclusion criteria for the MD-IBD part:

1. Male and female patients with IBD and 18 to 75 years of age.
2. Ability to understand and comply with the protocol.
3. Signed written Informed Consent.
4. Documented diagnosis of relapsing ileal, ileocolonic or colonic Crohn disease or relapsing ulcerative colitis.
5. Concomitant therapy (background medication) for inflammatory bowel disease: none or stable 8 weeks before baseline.
6. No signs of malignancy.

Exclusion criteria for the SAD and MAD part with healthy subjects:

1. Pre-existing relevant medical conditions.
2. Clinically relevant abnormal findings in medical history or screening assessments.
3. Participation in a clinical study.
4. Use of any prescribed or over-the-counter medication, food supplements or herbal preparations.
5. Use of antibiotics (systemic or gut-acting [non-absorbed]).
6. Pregnant or breastfeeding women or women of childbearing potential and male participants with female partners of childbearing age not using highly effective contraception till at least 1 month after last dosing of investigational medicinal product (IMP).
7. Legal incapacity.
8. Indications that the patient may be unable to comply with the study procedures, e.g. language barriers precluding adequate understanding or cooperation

Exclusion criteria for the MD-IBD part:

1. Diagnosis of indeterminate colitis, microscopic colitis, ischaemic colitis, infectious colitis, radiation colitis or diverticular disease (except for diverticles accompanying CD).
2. Current or past diagnosis of complex fistulae or intra-abdominal or peritoneal abscesses.
3. Strictures with obstructive symptoms.
4. Pregnant or breastfeeding women or women of childbearing potential and male participants with female partners of childbearing age not using highly effective contraception till at least 1 month after last dosing of investigational medicinal product (IMP).
5. Legal incapacity.
6. Indications that the patient may be unable to comply with the study procedures, e.g. language barriers precluding adequate understanding or cooperation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events [Safety and Tolerability] | up to 60 days
  Adverse Events (AEs) during treatment period
Treatment-Emergent Serious Adverse Events [Safety and Tolerability] | up to 60 days
  Serious Adverse Events (SAEs) during treatment period
Haemoglobin | up to 60 days
  Haemoglobin (Hb) in %
White blood cells | up to 60 days
  White blood cell (WBC) count as x10^9/l
Blood creatinine | up to 60 days
  Blood Creatinine in mmol/L
Blood urea | up to 60 days
  Urea in mmol/L
Blood uric acid | up to 60 days
  Uric acid in mmol/L
Glomerular filtration rate | up to 60 days
  Glomerular filtration rate (GFR, automatically calculated by the laboratory based on creatinine values) GFR in ml/min/1.73m2
Blood ALT | up to 60 days
  Alanine transaminase (ALT) in U/l
Blood AST | up to 60 days
  Aspartate transaminase (AST) in U/l
Blood GGT | up to 60 days
  Gamma glutamyl transferase (GGT) in U/l

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Nikolaus, Prof. Dr., Principal Investigator — University Medical Center Schleswig-Holstein, Campus Kiel
Locations (1):
- University Medical Center Schleswig-Holstein, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No